CLINICAL TRIAL: NCT03960476
Title: Decision Making and Implementation of Aging-in-Place/Long Term Care Plans Among Older Adults
Acronym: PYL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lee Lindquist, Associate Professor of Medicine, Section Chief - Geriatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AG058777 (NIH); 1R01AG058777-01A1 (NIH)
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Long-Term Care Planning
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: All study participants receive access to the web-based study intervention, PlanYourLifespan.org.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Access to Web-Based Intervention (Experimental): All study participants will be given access to the web-based study intervention, PlanYourLifespan.org.
  Interventions: Behavioral: PlanYourLifespan.org

INTERVENTIONS:
Behavioral: PlanYourLifespan.org — The study intervention is a web-based planning tool, PlanYourLifespan.org

SUMMARY:
This study seeks to better understand how older adult aging-in-place/long term care decision making and implementation is impacted by age-related changes (e.g. cognition, health literacy, chronic conditions) and social influences (e.g. caregivers/supporters).

DETAILED DESCRIPTION:
Subjects who are part of the National Institute on Aging (NIA)-funded LitCog study will be given access to PlanYourLifespan.org, a web-based decision-making and planning tool. Participants will be followed for up to 42 months to examine the mediating/moderating factors involved in decision-making, timing of decision implementation, and goal concordance. Findings have the potential to inform healthcare providers, caregivers, health/long term care insurers, area agencies on aging, and older adults nationally in supporting aging-in-place decisions and services use.

ELIGIBILITY:
Inclusion Criteria:

* Current participant in the LitCog Trial [R01AG03611]
* English-speaking
* Community-dwelling
* Currently use a computer or tablet with internet

Exclusion Criteria:

* Previous participation in the Advanced Planning for Home Services study [IH-12-11-4259]

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2026-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 293 Participants were recruited and given access to the web-based intervention PlanYourLifespan.org. Participants were assessed at Baseline, 1 month post baseline, and at 6 month intervals thereafter (6/12/18 months post baseline, etc). 36 Months Post-Baseline is the timepoint of interest for all primary and secondary outcomes. No partial data has been reported for any outcome. Reported data and values will not be updated.
Groups:
- All Enrolled Subjects: All study participants will be given access to the web-based study intervention, PlanYourLifespan.org.
Period: Baseline Assessment
Arm/Group | All Enrolled Subjects
Started | 293
Completed | 293
Not Completed | 0
Period: 1 month Assessment
Arm/Group | All Enrolled Subjects
Started | 293
Completed | 287
Not Completed | 6
Not completed — Unable to Contact | 4
Not completed — Subject Declined Assessment | 2
Period: 6 Month Assessment
Arm/Group | All Enrolled Subjects
Started | 293
Completed | 285
Not Completed | 8
Not completed — Death | 1
Not completed — Unable to Contact | 4
Not completed — Subject declined Assessment | 3
Period: 12 Month Assessment
Arm/Group | All Enrolled Subjects
Started | 292
Completed | 278
Not Completed | 14
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Unable to Contact | 8
Not completed — Subject Declined Assessment | 4
Period: 18 Month Assessment
Arm/Group | All Enrolled Subjects
Started | 290
Completed | 265
Not Completed | 25
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Unable to Contact | 19
Not completed — Subject Declined Assessment | 3
Period: 24 Month Assessment
Arm/Group | All Enrolled Subjects
Started | 287
Completed | 264
Not Completed | 23
Not completed — Death | 2
Not completed — Withdrawal by Subject | 4
Not completed — Unable to Contact | 10
Not completed — Subject Declined Assessment | 7
Period: 30 month assessment
Arm/Group | All Enrolled Subjects
Started | 281
Completed | 246
Not Completed | 35
Not completed — Withdrawal by Subject | 1
Not completed — Unable to contact | 22
Not completed — Subject declined Assessment | 12
Period: 36 Month Assessment
Arm/Group | All Enrolled Subjects
Started | 280
Completed | 240
Not Completed | 40
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Unable to Contact | 17
Not completed — Subject Declined Assessment | 17
Not completed — Participant Failed Pre-Assessment Cognition Testing | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 293
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Baseline
  years | 73.8 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex, Binary (Female/Male)
  Participants
    Female | 213
    Male | 80
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race (NIH/OMB)
  Participants
    American Indian or Alaska Native | 0
    Asian | 8
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 83
    White | 191
    More than one race | 3
    Unknown or Not Reported | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (NIH/OMB)
  Participants
    Hispanic or Latino | 13
    Not Hispanic or Latino | 273
    Unknown or Not Reported | 7
Rate of Participant Long-term care planning for Alzheimer's Dementia/Memory Loss [Count of Participants; unit: Participants] — Participants are asked 'If you developed Alzheimer's or memory loss and could no longer live independently in your home, have you decided what your living preferences (e.g. stay in own home, retirement/long term care community) would be?' Responses are recorded as binary (yes/no). Percentage below is percent of participants with an existing long term care plan at baseline.
  Participants | 121

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participant Long Term Care Planning for Alzheimer's Dementia/Memory Loss
Description: Participants were asked "If you developed Alzheimer's or memory loss and could no longer live independently in your home, have you decided what your living preferences (e.g. stay in own home, retirement/long term care community) would be?" Decision-making is measured as a binary ('yes', 'no') outcome at each time-point. Percentage given below is the % of participants who indicated "YES", that they have decided on their living preferences. All statistical analyses for this outcome reflect data at the 36 month assessment.
Time Frame: Assessed at baseline and every 6 months, 36 months reported
Population: 240 participants out of 293 had data available to report at 36 months Assessment. All participants with data available at 36 months post-baseline are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants | 173
Statistical Analysis 1: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing the fixed effect of marital status (unmarried) vs reference group (married), controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss. Corresponds to H2 in Protocol: Older adults with adequate social support will demonstrate a greater likelihood to complete decision-making for aging-in-place; Test type: Superiority; p = .6539, Mixed Models Analysis — Alpha for significance=0.05 for all tests; Odds Ratio (OR) = .966, 95% CI 2-sided [.66 to 1.414]
Statistical Analysis 2: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing the effect of Limited Health Literacy (vs adequate), as measured by the Newest Vital Sign index, controlling for repeated assessments within-subjects, on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss. Test corresponds to H4 in protocol: Older adults who have lower health literacy will be less likely to complete decision-making for aging-in-place; Test type: Superiority; p = .4178, Mixed Models Analysis — Alpha for significance=0.05 for all tests; Odds Ratio (OR) = .859, 95% CI 2-sided [.58 to 1.271]
Statistical Analysis 3: Comparison: All Enrolled Subjects; GLMM (all models evaluated in SAS 9.4) testing the effect of Limited Health Literacy (vs adequate), as measured by the Rapid Estimate of Adult Literacy in Medicine index, controlling for repeated assessments within-subjects, on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss.Test corresponds to H4 in protocol: Older adults who have lower health literacy will be less likely to complete decision-making for aging-in-place; Test type: Superiority; p = .7504, Mixed Models Analysis — Alpha for significance=0.05 for all tests; Odds Ratio (OR) = .704, 95% CI 2-sided [.405 to 1.224]
Statistical Analysis 4: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing the effect of former tobacco use (vs never used) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .9367, Mixed Models Analysis — alpha for significance p=0.05; Odds Ratio (OR) = 1.005, 95% CI 2-sided [.66 to 1.53]
Statistical Analysis 5: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing the effect of current tobacco use (vs never used) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .4337, Mixed Models Analysis; Odds Ratio (OR) = .745, 95% CI 2-sided [.29 to 1.914]
Statistical Analysis 6: Comparison: All Enrolled Subjects; GLMM (all models evaluated in SAS 9.4) testing level of Tangible Social Support (Adequate, vs ref no perceived need) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss. Test corresponds to H2. Older adults with adequate levels of social support will demonstrate a greater likelihood to complete decision-making for aging-in-place; Test type: Superiority; p = .0230, Mixed Models Analysis — alpha =0.05; Odds Ratio (OR) = 1.757, 95% CI 2-sided [.98 to 3.149]
Statistical Analysis 7: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing level of Tangible Social Support (more support needed, vs ref no perceived need) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .6664, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.361, 95% CI 2-sided [.782 to 2.371]
Statistical Analysis 8: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing affirmative use of the web-based intervention (Plan Your Lifespan tool, or PYL) in prior 12 months as a binary (yes/no) fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss. Corresponds to Protocol H3; Test type: Superiority; p = .6755, Mixed Models Analysis — alpha=.05; Odds Ratio (OR) = .975, 95% CI 2-sided [.732 to 1.297]
Statistical Analysis 9: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing for the effect of presence of cognitive impairment (any cognitive impairment=yes, vs reference group no) as fixed effect, controlling for repeated assessments within-subjects, on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .1228, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.295, 95% CI 2-sided [.827 to 2.028]
Statistical Analysis 10: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Consumer Health Activation- Low Activation (vs ref moderate activation) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .0438, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .779, 95% CI 2-sided [.510 to .802]
Statistical Analysis 11: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Consumer Health Activation- high Activation (vs ref moderate activation) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .5072, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.364, 95% CI 2-sided [.802 to 2.320]
Statistical Analysis 12: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Advance Care Planning- absence of a Living Will (vs ref level has living will) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .4130, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .916, 95% CI 2-sided [.652 to 1.288]
Statistical Analysis 13: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Advance Care Planning- does not have Power of Attorney (vs ref level has PoA) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .9268, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .827, 95% CI 2-sided [.594 to 1.153]
Statistical Analysis 14: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Event and Goal Concordance- No Hospitalization in past 6 months (vs ref level hospitalization prior 6 months) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .6247, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.222, 95% CI 2-sided [.817 to 1.828]
Statistical Analysis 15: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Event and Goal Concordance- New or Worsening Memory Loss in past 6 months (vs ref level no new/worsening Memory Loss, prior 6 months) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .9052, Mixed Models Analysis — Alpha=0.05; Odds Ratio (OR) = 1.052, 95% CI 2-sided [.68 to 1.628]
Statistical Analysis 16: Comparison: All Enrolled Subjects; GLMM in SAS 9.4 testing experiences with others- Hospitalization in past 6 months (vs ref level no experiences with others- hospitalization prior 6 months) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss. Participants were asked "In the past 6 months, have you had any personal experience with someone else who has been hospitalized?"; Test type: Superiority; p = .3663, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.060, 95% CI 2-sided [.836 to 1.344]
Statistical Analysis 17: Comparison: All Enrolled Subjects; GLMM in SAS 9.4 testing experiences with others- additional living support in past 6 months (vs ref level no experiences with others- additional living support) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for LTC in the event of ADML. Participants were asked "In the past 6 months, have you had any experiences with someone else requiring additional support in their home/needing to move into assisted living?"; Test type: Superiority; p = .8735, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.041, 95% CI 2-sided [.788 to 1.373]
Statistical Analysis 18: Comparison: All Enrolled Subjects; GLMM in SAS 9.4 testing experiences with others- any prior ADML experiences (vs ref level no prior ADML experiences with others) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for LTC in the event of ADML. Participants were asked "Have you had any prior experiences with someone else who has/ has had Alzheimer's disease and/or memory loss?"; Test type: Superiority; p = .1302, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.495, 95% CI 2-sided [1.143 to 1.954]
Statistical Analysis 19: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing age at baseline in years, continuous, as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .9337, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.013, 95% CI 2-sided [.976 to 1.052]
Statistical Analysis 20: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Months since Baseline, continuous, as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .0008, Mixed Models Analysis — alpha for significance=0.05; Odds Ratio (OR) = 1.047, 95% CI 2-sided [1.038 to 1.057]
Statistical Analysis 21: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Physical Function (measured by PROMIS Physical Function - Short Form 10a T score) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .0977, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.004, 95% CI 2-sided [.982 to 1.026]
Statistical Analysis 22: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Inductive Reasoning (measured by ETS Letter Sets score, ETS, 1976) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .8662, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .981, 95% CI 2-sided [.935 to 1.029]
Statistical Analysis 23: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Physical Function (measured by PROMIS Anxiety - Short Form 7a T score) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .6234, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.000, 95% CI 2-sided [.979 to 1.]
Statistical Analysis 24: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Working Memory (as measured by size judgment span index, cherry 1993) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .8307, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .993, 95% CI 2-sided [.833 to 1.184]
Statistical Analysis 25: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing subject processing speed (measured by digit comparison test, salthouse 1992) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .7311, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .988, 95% CI 2-sided [.974 to 1.003]
Statistical Analysis 26: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Long Term Memory (measured by New York Paragraph Test, Kruger 1999) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .634, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.01, 95% CI 2-sided [.951 to 1.073]
Statistical Analysis 27: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Depression (measured by PROMIS Depression- Short Form 8b T score) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .4889, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.005, 95% CI 2-sided [.983 to 1.027]
Statistical Analysis 28: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing subject Verbal Ability (measured by AM-NART score, Grober 1991) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .7556, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = .998, 95% CI 2-sided [.98 to 1.016]
Statistical Analysis 29: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Number of prescription medications, continuous, as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .8583, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.018, 95% CI 2-sided [.972 to 1.066]
Statistical Analysis 30: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Number of chronic conditions, continuous, as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .2647, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.066, 95% CI 2-sided [.960 to 1.185]
Statistical Analysis 31: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing subject Routinism levels, measured by the busyness and Routine Scale (Martin, 2003)as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .1253, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.068, 95% CI 2-sided [1 to 1.14]
Statistical Analysis 32: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing busyness, measured by the busyness and Routine Scale (Martin, 2003)as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .5368, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.008, 95% CI 2-sided [.969 to 1.047]
Statistical Analysis 33: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Subject Social Network Strength, measured by the Lubben Social Network Index ( Lubben 2006) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .4018, Mixed Models Analysis — alpha = 0.05; Odds Ratio (OR) = 1.013, 95% CI 2-sided [.979 to 1.049]
Statistical Analysis 34: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing General Self Efficacy (measured by PROMIS Self Efficacy T score) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .9930, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.000, 95% CI 2-sided [.984 to 1.016]
Statistical Analysis 35: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Self Efficacy in Social Interactions (measured by PROMIS Self Efficacy in Social Interactions- Short Form 4a T score) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .934, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1.005, 95% CI 2-sided [.988 to 1.022]
Statistical Analysis 36: Comparison: All Enrolled Subjects; Generalized Linear Mixed Model (all models evaluated in SAS 9.4) testing Subject Self- Management skills (measured by Curtis Comprehensive Health Activities Scale, Curtis 2015) as fixed effect, controlling for repeated assessments within-subjects, for the effect on the outcome of probability (OR) of planning for Long Term Care in the event of Alzheimer's Dementia/Memory Loss; Test type: Superiority; p = .9396, Mixed Models Analysis — alpha=0.05; Odds Ratio (OR) = 1, 95% CI 2-sided [.987 to 1.013]

2. Secondary Outcome: Rate of Participant Planning for In Home Care in the Event of Alzheimer's Disease/Memory Loss
Description: Participants were asked "Have you already decided what your preferences would be if you developed Alzheimer's Disease or memory loss and needed caregiver help in your home?". Responses recorded as binary. Percentage below is percentage of participants who reported positively that they had a plan for the scenario. Frequencies here are given for 36 month timepoint.
Time Frame: assessed 0-36 months, month 36 reported
Population: 240 Participants completed 36 Month Analysis and had available data to report.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants | 161

3. Secondary Outcome: Rate of Participant Planning for Memory Care in the Event of Alzheimer's Disease/Memory Loss
Description: Participants were asked "Have you decided what your long-term care preferences (e.g. where you would prefer to go if you needed to be in a nursing home or memory care), would be if you ever developed Alzheimer's Disease or memory loss? " Here, participants were specifically asked about "memory care" vs other types of care options. Responses recorded as binary. Percentage below is percentage of participants who reported positively ("Yes")that they had a plan for the scenario. Frequencies here are given for 36 month timepoint.
Time Frame: Assessed at 0-36 months, month 36 reported
Population: 240 Participants completed 36 Month Analysis and had available data to report.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants | 42

4. Secondary Outcome: Rate of Participant Planning for the Event of Hospitalization Requiring Rehabilitation Outside the Home
Description: Participants were asked "Have you already decided what your preferences would be if you were hospitalized and needed post-hospitalization rehabilitation outside of the home? " Responses recorded as binary. Percentage below is percentage of participants who reported positively ("Yes") that they had a plan for the scenario. Frequencies here are given for 36 month timepoint.
Time Frame: Assessed at 0-36 months, month 36 reported
Population: 240 Participants completed 36 Month Analysis and had available data to report.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants | 135

5. Secondary Outcome: Rate of Participant Planning for the Event of Hospitalization Requiring In-home Care
Description: Participants were asked "Have you already decided what your preferences would be if you were hospitalized and needed caregiver help in your home?" Responses recorded as binary. Percentage below is percentage of participants who reported positively ("Yes") that they had a plan for the scenario. Frequencies here are given for 36 month timepoint.
Time Frame: Assessed at 0-36 months, month 36 reported
Population: 240 Participants completed 36 Month Analysis and had available data to report.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants | 158

6. Secondary Outcome: Participant Decision Making Contemplation Rates- Alzheimer's Dementia/Memory Loss (ADML)
Description: Participants were asked a panel of statements about contemplation for decision-making in the event of Alzheimer's Dementia/Memory Loss (ADML). Participants were shown a statement and asked to gauge how frequently they contemplated the possibility of the given scenario, ranging from "Never" to "A lot". Frequencies given for 36 month timepoint per primary outcome analysis. Each statement is prefixed by "How much have you thought about..."
Time Frame: Assessed at 0-36 months, month 36 reported
Population: 240 participants had data available to report from 36 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: Never | 56
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: Once or Twice | 45
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: A Few Times | 41
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: Several Times | 21
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: A Lot | 31
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: N/A | 43
  How Alzheimer's Disease or memory loss could impact your ability to continue driving safely?: Unsure/Refused | 3
  How ADML might impact your ability to remain in your own home as you age?: Never | 41
  How ADML might impact your ability to remain in your own home as you age?: Once or Twice | 48
  How ADML might impact your ability to remain in your own home as you age?: A Few Times | 75
  How ADML might impact your ability to remain in your own home as you age?: Several Times | 41
  How ADML might impact your ability to remain in your own home as you age?: A Lot | 35
  How ADML might impact your ability to remain in your own home as you age?: N/A | 0
  How ADML might impact your ability to remain in your own home as you age?: Unsure/Refused | 0
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: Never | 50
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: Once or Twice | 56
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: A Few Times | 62
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: Several Times | 39
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: A Lot | 33
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: N/A | 0
  How ADML might require you to depend on an in-home caregiver (e.g. family member, paid caregiver)?: Unsure/Refused | 0
  How ADML might require you to use long-term care services (such as being in a nursing home)?: Never | 61
  How ADML might require you to use long-term care services (such as being in a nursing home)?: Once or Twice | 55
  How ADML might require you to use long-term care services (such as being in a nursing home)?: A Few Times | 60
  How ADML might require you to use long-term care services (such as being in a nursing home)?: Several Times | 36
  How ADML might require you to use long-term care services (such as being in a nursing home)?: A Lot | 28
  How ADML might require you to use long-term care services (such as being in a nursing home)?: N/A | 0
  How ADML might require you to use long-term care services (such as being in a nursing home)?: Unsure/Refused | 0
  The possibility of someone you love or know getting ADML in the future?: Never | 42
  The possibility of someone you love or know getting ADML in the future?: Once or Twice | 51
  The possibility of someone you love or know getting ADML in the future?: A Few Times | 66
  The possibility of someone you love or know getting ADML in the future?: Several Times | 55
  The possibility of someone you love or know getting ADML in the future?: A Lot | 26
  The possibility of someone you love or know getting ADML in the future?: N/A | 0
  The possibility of someone you love or know getting ADML in the future?: Unsure/Refused | 0
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: Never | 25
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: Once or Twice | 58
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: A Few Times | 80
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: Several Times | 50
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: A Lot | 27
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: N/A | 0
  Your possibility of getting Alzheimer's Disease or memory loss in the future?: Unsure/Refused | 0

7. Secondary Outcome: Participant Decision Making Contemplation Rates- Hospitalization
Description: Participants were asked a panel of statements about contemplation for decision-making in the event of Hospitalization. Participants were shown a statement and asked to gauge how frequently they contemplated the possibility of the given scenario, ranging from "Never" to "A lot". Frequencies given for 36 month timepoint per primary outcome analysis. Each statement is prefixed by "How much have you thought about..."
Time Frame: Assessed at 0-36 months, month 36 reported
Population: 240 participants had data available to report from 36 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants
  How a hospitalization could impact your ability to continue driving safely?: Never | 56
  How a hospitalization could impact your ability to continue driving safely?: Once or Twice | 53
  How a hospitalization could impact your ability to continue driving safely?: A Few Times | 43
  How a hospitalization could impact your ability to continue driving safely?: Several Times | 18
  How a hospitalization could impact your ability to continue driving safely?: A lot | 26
  How a hospitalization could impact your ability to continue driving safely?: N/A | 43
  How a hospitalization could impact your ability to continue driving safely?: Not Sure/Refused | 1
  How a hospitalization might impact your ability to remain in your own home as you age?: Never | 41
  How a hospitalization might impact your ability to remain in your own home as you age?: Once or Twice | 67
  How a hospitalization might impact your ability to remain in your own home as you age?: A Few Times | 59
  How a hospitalization might impact your ability to remain in your own home as you age?: Several Times | 34
  How a hospitalization might impact your ability to remain in your own home as you age?: A lot | 39
  How a hospitalization might impact your ability to remain in your own home as you age?: N/A | 0
  How a hospitalization might impact your ability to remain in your own home as you age?: Not Sure/Refused | 0
  How a hospitalization might require you to depend on an in-home caregiver?: Never | 36
  How a hospitalization might require you to depend on an in-home caregiver?: Once or Twice | 69
  How a hospitalization might require you to depend on an in-home caregiver?: A Few Times | 61
  How a hospitalization might require you to depend on an in-home caregiver?: Several Times | 30
  How a hospitalization might require you to depend on an in-home caregiver?: A lot | 44
  How a hospitalization might require you to depend on an in-home caregiver?: N/A | 0
  How a hospitalization might require you to depend on an in-home caregiver?: Not Sure/Refused | 0
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: Never | 69
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: Once or Twice | 62
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: A Few Times | 47
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: Several Times | 30
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: A lot | 32
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: N/A | 0
  How a hospitalization might require you to use long-term care services (such as a nursing home)?: Not Sure/Refused | 0
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: Never | 39
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: Once or Twice | 56
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: A Few Times | 65
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: Several Times | 35
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: A lot | 45
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: N/A | 0
  How a hospitalization might require you to use rehabilitation services (such as physical therapy)?: Not Sure/Refused | 0
  Possibly being hospitalized in the future?: Never | 41
  Possibly being hospitalized in the future?: Once or Twice | 59
  Possibly being hospitalized in the future?: A Few Times | 76
  Possibly being hospitalized in the future?: Several Times | 40
  Possibly being hospitalized in the future?: A lot | 24
  Possibly being hospitalized in the future?: N/A | 0
  Possibly being hospitalized in the future?: Not Sure/Refused | 0
  The possibility of someone you love or know being hospitalized in the future?: Never | 38
  The possibility of someone you love or know being hospitalized in the future?: Once or Twice | 68
  The possibility of someone you love or know being hospitalized in the future?: A Few Times | 73
  The possibility of someone you love or know being hospitalized in the future?: Several Times | 37
  The possibility of someone you love or know being hospitalized in the future?: A lot | 24
  The possibility of someone you love or know being hospitalized in the future?: N/A | 0
  The possibility of someone you love or know being hospitalized in the future?: Not Sure/Refused | 0

8. Secondary Outcome: Participant Utilization of Long-term Care Services
Description: Participant utilization of long-term care services such as in-home caregivers as measured by the Resource Use Inventory. Frequencies below are for "yes" responses to individual items on the inventory. This Outcome measure was only collected at the 18 month assessment time point and was collected as part of the LitCog assessment battery. Frequencies below reflect all available data at the 18 month assessment.
Time Frame: 18 month assessment
Population: 265 Participants completed the 18 month assessment point.
Measure: Count of Participants; unit: Participants
Arm/Group | Access to Web-Based Intervention
Number analyzed (Participants) | 265
Participants
  Has participant had any ambulatory surgeries or procedures in the past 12 months? | 87
  Has participant utilized ANY doctor (primary care, specialty or PT/OT) in the past 12 months? | 260
  Has participant had unpaid help with cleaning in the past 12 months? | 56
  Has participant utilized ANY medical equipment in the past 12 months? | 163
  Has participant visited Emergency Department in the past 12 months? | 66
  Has participant been admitted to a hospital in the past 12 months? | 37
  While admitted did participant have surgery?: number analyzed (Participants) | 37
  While admitted did participant have surgery? | 21
  After being discharged did participant utilize any post-hospital care?: number analyzed (Participants) | 37
  After being discharged did participant utilize any post-hospital care? | 7
  Has participant had unpaid help with laundry in the past 12 months? | 39
  Has participant had unpaid help with managing their money in the past 12 months? | 13
  Has participant had any form of unpaid help/care in the past 12 months? | 129
  Has participant utilized any paid help (help1) in the past 12 months? | 69
  Has participant been seen by a primary care provider in the past 12 months? | 238
  Has participant utilized physical or occupational therapy in the past 12 months? | 99
  Has participant utilized ANY scans in past year? | 184
  Has participant had unpaid help with shopping in the past 12 months? | 58
  Has participant seen ANY specialty care doctor in the past 12 months? | 216
  Has participant had unpaid help with transport in the past 12 months? | 91
  Has participant utilized urgent care in the past 12 months? | 79

9. Secondary Outcome: Previous Health Experiences- Self and Others
Description: Participants were asked a panel of non-validated questions about their previous health experiences and their experiences with others. Panel was collected at Baseline assessment only.
Time Frame: Baseline
Population: Only Participants reporting hospitalization were asked follow-up question about post-hospitalization rehabilitation. Only Participants reporting memory loss were asked follow up question. Only participants reporting prior experience with others with memory loss were asked follow up question.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 293
Participants
  In the Past 3 Years, have you been hospitalized?: No | 190
  In the Past 3 Years, have you been hospitalized?: Yes | 99
  In the Past 3 Years, have you been hospitalized?: Unsure/Don't Know | 4
  Did you need assistance or therapy after your hospitalization?: number analyzed (Participants) | 99
  Did you need assistance or therapy after your hospitalization?: No | 48
  Did you need assistance or therapy after your hospitalization?: Yes | 51
  Did you need assistance or therapy after your hospitalization?: Unsure/Don't Know | 0
  Have you had any prior personal experience with someone who has been hospitalized?: No | 51
  Have you had any prior personal experience with someone who has been hospitalized?: Yes | 242
  Have you had any prior personal experience with someone who has been hospitalized?: Unsure/Don't Know | 0
  Have you had any prior experiences with someonerequiring additional support in their home?: No | 107
  Have you had any prior experiences with someonerequiring additional support in their home?: Yes | 185
  Have you had any prior experiences with someonerequiring additional support in their home?: Unsure/Don't Know | 1
  Have you had any prior experience with someone needing to move into a supportive living environment?: No | 138
  Have you had any prior experience with someone needing to move into a supportive living environment?: Yes | 153
  Have you had any prior experience with someone needing to move into a supportive living environment?: Unsure/Don't Know | 2
  Have you experienced any memory loss?: No | 144
  Have you experienced any memory loss?: Yes | 139
  Have you experienced any memory loss?: Unsure/Don't Know | 10
  Do you feel that this memory loss is normal for your age?: number analyzed (Participants) | 139
  Do you feel that this memory loss is normal for your age?: No | 13
  Do you feel that this memory loss is normal for your age?: Yes | 109
  Do you feel that this memory loss is normal for your age?: Unsure/Don't Know | 17
  Have you had prior experience with someone else who has/had Alzheimer's disease and/or memory loss?: No | 81
  Have you had prior experience with someone else who has/had Alzheimer's disease and/or memory loss?: Yes | 212
  Have you had prior experience with someone else who has/had Alzheimer's disease and/or memory loss?: Unsure/Don't Know | 0
  Did they require any help or assistance due to their condition?: number analyzed (Participants) | 212
  Did they require any help or assistance due to their condition?: No | 18
  Did they require any help or assistance due to their condition?: Yes | 181
  Did they require any help or assistance due to their condition?: Unsure/Don't Know | 13

10. Other Pre Specified Outcome: Website Satisfaction Assessment
Description: Participants assessed their satisfaction with the PlanYourLifespan.org website tool after use at Baseline. Participants ranked agreement with 8 statements regarding website utilization and satisfaction on a 1-5 point likert scale with values ranging from "strongly agree" to "strongly disagree".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 293
Participants
  This website is easy to use.: Strongly Agree | 119
  This website is easy to use.: Agree | 147
  This website is easy to use.: Neutral or Unsure | 20
  This website is easy to use.: Disagree | 5
  This website is easy to use.: Strongly Disagree | 1
  This website is easy to use.: Prefer not to say/Refused | 1
  Terminology used on this website is clear.: Strongly Agree | 123
  Terminology used on this website is clear.: Agree | 165
  Terminology used on this website is clear.: Neutral or Unsure | 5
  Terminology used on this website is clear.: Disagree | 0
  Terminology used on this website is clear.: Strongly Disagree | 0
  Terminology used on this website is clear.: Prefer not to say/Refused | 0
  The content on this website met my expectations.: Strongly Agree | 77
  The content on this website met my expectations.: Agree | 150
  The content on this website met my expectations.: Neutral or Unsure | 57
  The content on this website met my expectations.: Disagree | 3
  The content on this website met my expectations.: Strongly Disagree | 3
  The content on this website met my expectations.: Prefer not to say/Refused | 3
  This website is visually appealing.: Strongly Agree | 81
  This website is visually appealing.: Agree | 164
  This website is visually appealing.: Neutral or Unsure | 38
  This website is visually appealing.: Disagree | 9
  This website is visually appealing.: Strongly Disagree | 0
  This website is visually appealing.: Prefer not to say/Refused | 1
  It was easy to move from one page to the next.: Strongly Agree | 113
  It was easy to move from one page to the next.: Agree | 155
  It was easy to move from one page to the next.: Neutral or Unsure | 16
  It was easy to move from one page to the next.: Disagree | 9
  It was easy to move from one page to the next.: Strongly Disagree | 0
  It was easy to move from one page to the next.: Prefer not to say/Refused | 0
  I was able to complete my tasks on the website in a reasonable amount of time.: Strongly Agree | 79
  I was able to complete my tasks on the website in a reasonable amount of time.: Agree | 173
  I was able to complete my tasks on the website in a reasonable amount of time.: Neutral or Unsure | 26
  I was able to complete my tasks on the website in a reasonable amount of time.: Disagree | 10
  I was able to complete my tasks on the website in a reasonable amount of time.: Strongly Disagree | 3
  I was able to complete my tasks on the website in a reasonable amount of time.: Prefer not to say/Refused | 2
  I would be likely to use this website in the future.: Strongly Agree | 90
  I would be likely to use this website in the future.: Agree | 149
  I would be likely to use this website in the future.: Neutral or Unsure | 38
  I would be likely to use this website in the future.: Disagree | 15
  I would be likely to use this website in the future.: Strongly Disagree | 1
  I would be likely to use this website in the future.: Prefer not to say/Refused | 0
  I would recommend this website to others.: Strongly Agree | 96
  I would recommend this website to others.: Agree | 154
  I would recommend this website to others.: Neutral or Unsure | 33
  I would recommend this website to others.: Disagree | 10
  I would recommend this website to others.: Strongly Disagree | 0
  I would recommend this website to others.: Prefer not to say/Refused | 0

11. Secondary Outcome: Event and Goal Concordance
Description: Participants are assessed at each timepoint regarding hospitalization events, recent memory loss, and changes in lifestyle due to hospitalization and memory loss. Responses are binary (yes/no), with a N/A and "unsure/don't know" option. Questions are non-validated. Frequencies given here are from 36 Month timepoint.
Time Frame: Assessed at 0-36 months, month 36 reported
Population: 240 Participants had data available at the 36 month timepoint. Follow-up questions regarding hospitalization were only deployed to participants who indicated a hospitalization event in the prior six months (n=36). Follow-up questions regarding memory loss were only deployed to participants who indicated new or worsening memory loss in the prior six months (n=42).
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 240
Participants
  In the past 6 months have you been hospitalized?: No | 204
  In the past 6 months have you been hospitalized?: Yes | 36
  In the past 6 months have you been hospitalized?: N/A | 0
  In the past 6 months have you been hospitalized?: Not Sure/Don't Know | 0
  Did you need any therapy/rehabilitation after any of your hospitalizations?: number analyzed (Participants) | 36
  Did you need any therapy/rehabilitation after any of your hospitalizations?: No | 21
  Did you need any therapy/rehabilitation after any of your hospitalizations?: Yes | 15
  Did you need any therapy/rehabilitation after any of your hospitalizations?: N/A | 0
  Did you need any therapy/rehabilitation after any of your hospitalizations?: Not Sure/Don't Know | 0
  Did you need any help in your home after any of your hospitalizations?: number analyzed (Participants) | 36
  Did you need any help in your home after any of your hospitalizations?: No | 24
  Did you need any help in your home after any of your hospitalizations?: Yes | 12
  Did you need any help in your home after any of your hospitalizations?: N/A | 0
  Did you need any help in your home after any of your hospitalizations?: Not Sure/Don't Know | 0
  In the past 6 months, have you experienced any new or worsening memory loss?: No | 196
  In the past 6 months, have you experienced any new or worsening memory loss?: Yes | 42
  In the past 6 months, have you experienced any new or worsening memory loss?: N/A | 0
  In the past 6 months, have you experienced any new or worsening memory loss?: Not Sure/Don't Know | 2
  Do you think memory loss is normal for your age?: number analyzed (Participants) | 42
  Do you think memory loss is normal for your age?: No | 7
  Do you think memory loss is normal for your age?: Yes | 31
  Do you think memory loss is normal for your age?: N/A | 0
  Do you think memory loss is normal for your age?: Not Sure/Don't Know | 4
  Did your memory loss affect where you currently live/did you make any physical changes to your home?: number analyzed (Participants) | 42
  Did your memory loss affect where you currently live/did you make any physical changes to your home?: No | 42
  Did your memory loss affect where you currently live/did you make any physical changes to your home?: Yes | 0
  Did your memory loss affect where you currently live/did you make any physical changes to your home?: N/A | 0
  Did your memory loss affect where you currently live/did you make any physical changes to your home?: Not Sure/Don't Know | 0
  Did your experience(s) with memory loss in the past 6 months affect your driving?: number analyzed (Participants) | 42
  Did your experience(s) with memory loss in the past 6 months affect your driving?: No | 26
  Did your experience(s) with memory loss in the past 6 months affect your driving?: Yes | 2
  Did your experience(s) with memory loss in the past 6 months affect your driving?: N/A | 13
  Did your experience(s) with memory loss in the past 6 months affect your driving?: Not Sure/Don't Know | 1
  Did your experience(s) with memory loss make you need any in-home caregiver assistance?: number analyzed (Participants) | 42
  Did your experience(s) with memory loss make you need any in-home caregiver assistance?: No | 40
  Did your experience(s) with memory loss make you need any in-home caregiver assistance?: Yes | 2
  Did your experience(s) with memory loss make you need any in-home caregiver assistance?: N/A | 0
  Did your experience(s) with memory loss make you need any in-home caregiver assistance?: Not Sure/Don't Know | 0

ADVERSE EVENTS:
Time Frame: From Enrollment until end of follow-up, 36 months post-baseline
Description: SAEs (inpatient psychiatry admissions, worsening depression, hospitalization due to emotional reasons) AEs (increased emotional stress, increased anxiety over decision making, increased anxiety with communication plans with relatives and surrogates, increased conflict with relatives over communicating decisions)
  All-Cause Mortality Rate below reflects all deaths reported from Baseline-36 month assessment period.
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 7/293
Serious Adverse Events (participants affected / at risk) | 0/293
Other Adverse Events (participants affected / at risk) | 0/293

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03960476/Prot_SAP_000.pdf